CLINICAL TRIAL: NCT04090060
Title: Determining the Accuracy of Self and Partner Anal Exams for Detecting Anal Abnormalities.
Brief Title: The Prevent Anal Cancer Palpation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Chicago (Other); M.D. Anderson Cancer Center (Other); The University of Texas Health Science Center, Houston (Other); Gordon Crofoot MD PA (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alan Nyitray, PhD, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PRO00033000; R01CA232892-01 (NIH)
Record Dates: First submitted 2019-09-05; First posted 2019-09-16 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Anal Cancer
Keywords: Anus neoplasm; Digital anal rectal examination; Self anal examination
MeSH Terms: conditions — Anus Neoplasms

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to groups encouraged to practice anal examination (Experimental) or not encouraged to practice anal examinations (Control).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Practice Self-/Companion Exams (Experimental): 300 individuals and 50 couples will be randomized to practice arm.
  Interventions: Behavioral: Practice Self-/Companion Exams
- Control Arm (Other): 300 individuals and 50 couples will neither be encouraged nor discouraged to practice self-/companion exam.
  Interventions: Behavioral: Control Arm

INTERVENTIONS:
Behavioral: Practice Self-/Companion Exams — 300 men and 50 couples will be randomized and encouraged to practice anal exams at home before Visit 2. Practice results will be elicited by staff. They will return for Visit 2 (six months after Visit 1). At Visit 2, they will complete a pre- and post-visit computer assisted self-interview. They will receive written instructions. After completing an anal self-exam or anal companion exam at home, they will record the results. At the clinic, they will have a Digital Anal Rectal Exam (DARE) by a clinician who will give the subject his results.
  Arms: Practice Self-/Companion Exams
Behavioral: Control Arm — 300 individuals and 50 couples will be randomized to this arm. Following Visit 1, they will neither be encouraged nor discouraged from practicing self- or companion exam. They will return for Visit 2 (six months after Visit 1). They will receive written anal exam instructions. They will then complete the self- or companion exam at home, and record the results. At the clinic, they will receive a clinician DARE. Clinicians will give DARE results. Persons will take a post-exam computer-assisted self-interview. Persons in this arm (control) will be asked if they have performed exams between visits.
  Arms: Control Arm

SUMMARY:
Anal cancer is a common cancer among men having sex with men (MSM). We will investigate increasing detection of anal canal tumors through self- or partner-palpation of the anal canal among MSM and trans persons. This study in Houston and Chicago will recruit a sample of 100 couples (i.e., 200 partners) and 600 single persons (one-half HIV-positive), aged ≥ 25 years, who will be taught to perform an ASE or ACE. After performing the exam in private, the individual's ASE and partner's ACE will then be compared with a clinician's DARE. The assessment will be done at each of two visits, spaced 6-months apart. One-half of persons will be randomized to a practice condition to assess how practice affects accuracy and retention of exam procedure. Our hypothesis is that both ASE and ACE at visit 1 will have ≥70% sensitivity and ≥90% specificity using the clinician DARE as the gold standard at each of two visits.

DETAILED DESCRIPTION:
Even though expert opinion recommends annual digital ano-rectal exams (DARE) for detection of anal cancer tumors among men having sex with men (MSM), the procedure is severely underutilized by clinicians and it is not known how to increase utilization. This is problematic in the context of an extremely high incidence of anal cancer among MSM, no proven treatment for anal precancerous lesions, and lack of screening infrastructure for detecting precancerous lesions, even in high-resource countries.

The long-term goal of this study is to decrease morbidity and mortality from anal cancer by increasing detection of anal canal tumors through self- or partner-palpation of the anal canal. Preliminary data indicate these exams are feasible and highly acceptable among MSM. In a diverse sample of 200 MSM, 93% of men correctly classified their anal self-exam (ASE) or anal companion exam (ACE) as either normal or abnormal, and 94% said the exams were acceptable. Given these findings, our overall objective is to determine the viability of the ASE and ACE by assessing exam accuracy and consistency of results in two clinic sites. Accuracy will be defined as concordance between clinician DARE and participant exam. The central hypothesis is that both ASE and ACE at visit 1 will have ≥70% sensitivity and ≥90% specificity using the clinician DARE as the gold standard at each of two visits. We will test the hypothesis with three specific aims: 1) Estimate ASE and ACE sensitivity and specificity; 2) Determine independent factors associated with ASE and ACE concordance; and 3) Determine the impact of ASE, ACE, and DARE on survival and quality of life, and evaluate the cost-effectiveness of these strategies among HIV+ and HIV- MSM and transgender persons. The aims will be accomplished with a study in Houston and Chicago with a sample of 100 couples (i.e., 200 partners) and 600 single persons (one-half HIV-positive), aged >=25 years, who will perform a clinician-taught ASE or ACE. The individual's ASE and partner's ACE will then be compared with the clinician's DARE. The assessment will be done at each of two visits, spaced six-months apart, to assess retention of exam accuracy.

At the end of visit 1, one-half of participants, i.e., 300 individuals and 50 couples (stratified by city) will be randomly selected and encouraged to practice the ASE/ACE three months before Visit 2. Study staff will make reminder calls (or emails/texts) and follow-up calls for the scheduled practice session. At the follow-up calls, study staff will record the participant's result for the self/companion exam and the level of anxiety and pain, if any, associated with the exam. If the participant reports more than minimal pain and anxiety, they will be asked to return to the clinic for an exam. Regardless of prior results, all persons will be asked to return for Visit 2.

ELIGIBILITY:
Inclusion Criteria:

* Chicago or Houston Metro Residents
* Persons who had sex with men in the prior five years
* Cis-gendered men and transgender persons
* Age: 25 years and over
* Access to medical care for referral or treatment
* Spanish or English speakers/readers
* Individuals or couples
* HIV+ or HIV-
* Persons with or without comorbidities and physical disabilities

Exclusion Criteria:

* Unresolved health care provider's diagnosis of anal condyloma, hemorrhoids or anal cancer
* DARE in the prior three months
* Plans to move in the following six months

Min Age: 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cis-gendered men and transgender persons.
Enrollment: 718 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Nyitray, PhD, Principal Investigator — Medical College of Wisconsin
Locations (4):
- United States (4):
  - University of Chicago, Chicago, Illinois
  - Medical University of South Carolina, Charleston, South Carolina
  - M.D. Anderson Cancer Center, Houston, Texas
  - Gordon Crofoot MD, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nyitray AG, Rosser BRS, Hazra A, Nitkowski J, Smith D, Brzezinski B, Ridolfi TJ, Schneider JA, Chiao EY, Sanos S, Mkonyi E, Mgopa L, Ross MW. Factors associated with decreased anal sphincter tone and the accuracy of forced anal examinations to detect individuals having receptive anal intercourse: an observational study. BMJ Public Health. 2024 Jul 12;2(1):e001039. doi: 10.1136/bmjph-2024-001039. eCollection 2024 Jun. PMID 40018098
- [Derived] Nyitray AG, Rosser BRS, Hazra A, Nitkowski J, Smith D, Brzezinski B, Ridolfi TJ, Schneider JA, Chiao EY, Sanos S, Mkonyi E, Mgopa LR, Ross MW. Factors associated with decreased anal sphincter tone and the accuracy of forced anal examinations to detect individuals having receptive anal intercourse: An observational study. medRxiv [Preprint]. 2024 Feb 1:2024.01.31.24302098. doi: 10.1101/2024.01.31.24302098. PMID 38352524

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After consenting online, individuals must have attended a visit 1 where the intervention was delivered and followed by randomization into Practice or Control arms. The stated number of enrollees, 718, represents unique individuals who attended visit 1 and received the intervention regardless of the individual choosing to participate in the intervention as a single person or with a partner. The outcomes are assessed at the individual level and not couple level.
Groups:
- Practice Self-/Companion Exams: 300 individuals and 50 couples will be randomized to practice arm.
  Practice Self-/Companion Exams: 300 men and 50 couples will be randomized and encouraged to practice anal exams at home before Visit 2. Practice results will be elicited by staff. They will return for Visit 2 (six months after Visit 1). At Visit 2, they will complete a pre- and post-visit computer assisted self-interview. They will receive written instructions. After completing an anal self-exam or anal companion exam at home, they will record the results. At the clinic, they will have a Digital Anal Rectal Exam (DARE) by a clinician who will give the subject his results.
  Thus the Overall Number of Baseline Participants, Overall number of Participants Analyzed and Number of Participants at Risk reflect a unique number of participants and NOT a combination of participants and dyads.
- Control Arm: 300 individuals and 50 couples will neither be encouraged nor discouraged to practice self-/companion exam.
  Control Arm: 300 individuals and 50 couples will be randomized to this arm. Following Visit 1, they will neither be encouraged nor discouraged from practicing self- or companion exam. They will return for Visit 2 (six months after Visit 1). They will receive written anal exam instructions. They will then complete the self- or companion exam at home, and record the results. At the clinic, they will receive a clinician DARE. Clinicians will give DARE results. Persons will take a post-exam computer-assisted self-interview. Persons in this arm (control) will be asked if they have performed exams between visits.
  The Overall Number of Baseline Participants, Overall number of Participants Analyzed and Number of Participants at Risk reflect a unique number of participants and NOT a combination of participants and dyads.
Period: Overall Study
Arm/Group | Practice Self-/Companion Exams | Control Arm
Started | 359 | 359
Completed | 283 | 282
Not Completed | 76 | 77
Not completed — Lost to Follow-up | 76 | 77

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Practice Self-/Companion Exams | Control Arm | Total
Number analyzed (Participants) | 359 | 359 | 718
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 340 | 342 | 682
  >=65 years | 19 | 17 | 36
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 337 | 338 | 675
  Female | 1 | 0 | 1
  Trans Man | 3 | 6 | 9
  Trans Woman | 7 | 4 | 11
  Non-Binary | 10 | 8 | 18
  Other | 1 | 2 | 3
  Not Reported | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 92 | 72 | 164
  Not Hispanic or Latino | 266 | 286 | 552
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 4 | 13
  Asian | 11 | 22 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 88 | 93 | 181
  White | 217 | 212 | 429
  More than one race | 30 | 20 | 50
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 359 | 359 | 718

OUTCOME MEASURES:

1. Primary Outcome: Concordance Between Self-examination and Clinician Examination
Description: This measure will record the number of concordant digital anal examination results. A concordant result means that the subject and clinician agree as to the presence or absence of an abnormality.
Time Frame: Day 1
Population: Of 718 individuals, outcome results were available for 714 individuals with two participants in the Practice Self/Companion Exams arm and two participants in the Control Arm not completing the self-/companion examination or not completing a digital anal rectal examination. Of the 714, 357 were in the practice arm and 357 in the control arm. Of the 714, 658 completed a self-exam and 56 completed a companion exam.
Measure: Count of Participants; unit: Participants
Groups:
- Practice Self-/Companion Exams: 300 individuals and 50 couples will be randomized to practice arm.
  Practice Self-/Companion Exams: 300 individuals and 50 couples will be randomized and encouraged to practice anal exams at home before Visit 2. Practice results will be elicited by staff. They will return for Visit 2 (six months after Visit 1). At Visit 2, they will complete a pre- and post-visit computer assisted self-interview. They will receive written instructions. After completing an anal self-exam or anal companion exam at home, they will record the results. At the clinic, they will have a Digital Anal Rectal Exam (DARE) by a clinician who will give the subject his results.
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 331 | 327
Participants | 234 | 247

2. Primary Outcome: Concordance Between Self-examination and Clinician Examination
Description: as for outcome 1
Time Frame: Day 180.
Population: Seventy of 331 participants in the Practice Self-Companion Exams arm and 72 of 327 participants in the control arm completing a baseline examination (Outcome Measure 1) did not complete an examination at 180 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 261 | 255
Participants | 248 | 246

3. Primary Outcome: Concordance Between Companion Examination and Clinician Examination
Description: This measure will record the number of concordant digital anal examination results. A concordant result means that the subject's companion and clinician agree as to the presence or absence of an abnormality.
Time Frame: Day 1
Population: The unit of analysis is the individual and not the couple.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 26 | 30
Participants | 20 | 22

4. Primary Outcome: Concordance Between Companion Examination and Clinician Examination
Description: as for outcome 3
Time Frame: Day 180
Population: Twenty of twenty-six participants in the Practice Self-/Companion Exams arm and twenty-six of thirty participants in the Control Arm completed companion examinations at 180 days.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 20 | 26
Participants | 19 | 23

5. Primary Outcome: Number of Persons Who Practice the Self Examination
Description: This measure will count the number of subjects who practiced the self examination at least one time between days 1 and 180.
Time Frame: Day 180
Population: All units of data are unique individuals and not couples.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 331 | 327
Participants | 261 | 255

6. Primary Outcome: Number of Persons Who Practice the Companion Examination
Description: This measure will count the number of subjects who practiced the companion examination at least one time between days 1 and 180.
Time Frame: Day 180
Population: The unit of analysis is the individual not the dyad (or couple).
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 26 | 30
Participants | 20 | 26

7. Secondary Outcome: Measuring the Difference Between Chicago and Houston Self-exam Concordance.
Description: This measure will count the number of subjects in outcome measures 1, 2, 5 and 9 comparing subjects living in the Chicago and Houston metropolitan areas.
Time Frame: Day 1
Population: This measure involves only the participants living in either the Chicago or Houston metropolitan areas.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 331 | 327
Participants
  Chicago: number analyzed (Participants) | 177 | 175
  Chicago | 127 | 139
  Houston: number analyzed (Participants) | 154 | 152
  Houston | 107 | 108

8. Secondary Outcome: Measuring the Difference Between Chicago and Houston Companion Exam Concordance.
Description: This measure will count the number of subjects in outcome measures 3, 4, 6 and 9 comparing companions living in the Chicago and Houston metropolitan areas.
Time Frame: Day 1
Population: This measure involves only the participants living in either the Chicago or Houston metropolitan areas who conducted companion examinations.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 26 | 30
Participants
  Chicago: number analyzed (Participants) | 10 | 8
  Chicago | 10 | 6
  Houston: number analyzed (Participants) | 16 | 22
  Houston | 10 | 16

9. Secondary Outcome: Waist Circumference for Persons Doing Self-examinations
Description: This measure will record subject waist circumference in cm.
Time Frame: Day 1
Population: Waist circumference was not measured for 2 individuals in the practice arm and 2 individuals in the control arm.
Measure: Median (Full Range); unit: centimeter
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 329 | 325
centimeter | 96.1 [66.0 to 171.2] | 95.3 [66.6 to 178.0]

10. Secondary Outcome: Concordance Between Self-examination and Clinician Examination Stratified by Waist Circumference.
Description: This measure will record the number of concordant digital anal examination results in persons with less than or equal to 102 cm waist size versus greater than 102 cm waist size. A concordant result means that the subject and clinician agree as to the presence or absence of an abnormality.
Time Frame: Day 1
Population: This measure involves only the participants who performed a self-examination and whose waste circumference was measured. Two participants in each arm were missing waist circumference.
Measure: Count of Participants; unit: Participants
Arm/Group | Practice Self-/Companion Exams | Control Arm
Number analyzed (Participants) | 329 | 325
Participants
  Circumference <= 102 cm: number analyzed (Participants) | 214 | 222
  Circumference <= 102 cm | 153 | 174
  Circumference >102 cm: number analyzed (Participants) | 115 | 103
  Circumference >102 cm | 79 | 71

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Practice Self-/Companion Exams | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/359 | 0/359
Serious Adverse Events (participants affected / at risk) | 0/359 | 0/359
Other Adverse Events (participants affected / at risk) | 0/359 | 0/359

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-20): https://cdn.clinicaltrials.gov/large-docs/60/NCT04090060/Prot_SAP_002.pdf
  • Informed Consent Form (2022-05-15): https://cdn.clinicaltrials.gov/large-docs/60/NCT04090060/ICF_001.pdf